CLINICAL TRIAL: NCT03588767
Title: Endocrine Response of the Organism to Polytrauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCP-UP-TRAUMA; RVO-FNO/2017 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2018-06-26; First posted 2018-07-17 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Polytrauma
Keywords: polytrauma; endocrine response; metabolic response; bone metabolism; anabolic substance; vitamin D
MeSH Terms: conditions — Multiple Trauma | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Patients with polytrauma will be administered vitamin D3 + anabolic substance. Group of an identical size of patients who were treated in the past without administration of vitamin D3 and anabolic substance will be analyzed retrospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 + anabolic substance (Experimental): Prospectively enrolled patients with polytrauma, administration of vitamin D3 + anabolic substance
  Interventions: Drug: Vitamin D3 + anabolic substance
- Retrospective analysis (Active Comparator): Retrospectively analyzed patients, no vitamin D3 + anabolic substance administration.
  Interventions: Other: No Vitamin D3 + anabolic substance

INTERVENTIONS:
Drug: Vitamin D3 + anabolic substance — Prospectively enrolled patients with polytrauma, administration of vitamin D3 + anabolic substance
  Arms: Vitamin D3 + anabolic substance
Other: No Vitamin D3 + anabolic substance — Retrospectively analyzed group of patients, no Vitamin D3 + anabolic substance administration
  Arms: Retrospective analysis

SUMMARY:
The serious injury causes a complex acute response of the organism to the injury in affected patients, which is manifested in the neuroendocrine, immune and metabolic areas, with an often persisting catabolic state, with a subsequent negative impact upon bone metabolism.

By a timely administration of the D3 vitamin and an anabolic, we attempt to achieve an earlier activation of the anabolic phase of patient resuscitation after serious trauma regarding the monitoring of laboratory values of bone metabolism.

DETAILED DESCRIPTION:
Polytrauma and serious complex injuries evoke a vast acute response of the organism to the injury in patients with serious trauma, not only in the form of trauma-haemorrhagic instability; the metabolic response of the organism to trauma also changes, these changes are manifested with activation of integration systems, in the areas of hemocoagulation, as well as changes in the form of changes in the endocrine and immunology systems. The extent of these changes always depends upon the extent and intensity of the mechanism of injury, together with the extent and type of impairment of individual organ systems in the polytraumatized patient.

1. primarily, due to the extent of the anatomic injury caused by trauma
2. due to the need to mobilize the reserves in order to repair the impaired tissues
3. due to the need to activate the main integration systems in the following areas: endocrine, neurological and immunology

Immediately after the injury, the organism reacts to the load with acute phase response, which is characterized with stimulation of the hypothalamus-hypophysis-adrenal glands axis, with activation of the sympathoadrenal system, furthermore with stimulation of synthesis of proteins of the acute phase, activation of the immune system (B-cells and T-cells), activation of neutrophils, fibroblasts, and endothelial cells. At the same time, significant catabolism of proteins occurs, together with changes of levels of various hormones. This pertains primarily to an early decrease of levels of anabolic-acting testosterone, dihydrotestosterone, and free testosterone, and also the total and ionized calcium, high levels of the parathyroid hormone, interleukin-6, cortisol and changes in thyroidal hormones, etc.

At present, substation therapy with an early administration of a substitution dose of vitamin D3 after determination of its level is recommended to treat this endocrine reaction, together with anabolic substances, such as nandrolone decanoate (Deca-Durabolin) already on the first day, while respecting the contraindications, with the aim to reverse the catabolic phase of the polytrauma into the anabolic phase, which, apart from other indicators, influences the parameters of bone metabolism, which may be monitored in the laboratory.

The aim of the study is to verify, whether the administration of substitution vitamin D3 does and anabolic-acting Deca-Durabolin substance (concomitant) from the beginning of the treatment leads to

1. elimination of bone reabsorption
2. earlier initiation of the bone remodeling phase in patients affected with a polytrauma, in comparison with a group of similarly traumatized patients from a retrospective file, who did not receive this treatment.

A group of 30 polytraumatized patients with administration of vitamin D3 and Deca-Durabolin anabolic substance will be retrospectively compared to a group of patients treated at the Department of Trauma Surgery, University Hospital Ostrava with ISS>31 in the past years.

Administered substances

1. Vitamin D3 - Bon 200 000 I.U. i.m. on the first day of trauma, and 3 weeks after trauma, following the verification of 25/OH/ vitamin D value, further substitution of vitamin D in the form of Vigantol 5000I.U. drops administered per os once a week for the period of 6 weeks; the total period of treatment lasting 9 weeks
2. Anabolic substance - Deca-Durabolin 50mg i.m. on the first day of trauma, a repeated dose of Deca-Durabolin 50mg i.m. 1amp. every 3 weeks; the total period of treatment lasting 9 weeks

Parameters of the bone metabolism and endocrine response will be monitored (telopeptide CTx- beta mass, bone alkaline phosphatase, osteocalcin, type-I procollagen propeptide, bone fraction of alkaline phosphatase, total and ionized calcium, S+U, phosphorus S+U, parathyroid hormone, 25-OH vitamin D, Cortisol S+U , testosterone, dihydrotestosterone, free testosterone, T3, fT4, 17 beta-estradiol/, interleukin 6. These parameters were monitored on the 1st, 7th, 14th, 28th and 70th day.

The results will be analyzed with statistical methods for the purpose of further assessment and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* serious polytrauma with ISS>31b
* females, 18-50 years of age
* males, 18-60 years of age
* signed informed consent with participation in the study

Exclusion Criteria:

* infaust craniocerebral injury
* gravidity
* lactation
* prostate cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Different age limits in males and females will be used as eligibility criteria for patients enrolled in the study. Males of 18-60 years of age and females of 18-50 years of age will be eligible for participation in the study. This difference is explained by the different bone metabolism in male and female patients.
Enrollment: 60 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Bone metabolism | 39 months
  Measurement of the P1NP parameter of bone metabolism (earlier bone remodelling): increase of the P1NP parameter over 170% on the 70th day after injury - yes/no

SECONDARY OUTCOMES:
Time of healing in patients with multiple fractures | 39 months
  The time of healing will be assessed in patients with multiple fractures - measured in the number of months until complete healing is confirmed with radio diagnostic examination (X-ray)

CONTACTS AND LOCATIONS:
Overall Officials: Renáta Ječmínková, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data my be provided upon request.